CLINICAL TRIAL: NCT03508661
Title: The Scleroderma Patient-centered Intervention Network (SPIN) - Scleroderma Support Group Leader EDucation (SSLED) Program Feasibility Trial
Brief Title: The Scleroderma Patient-centered Intervention Network (SPIN) Support Group Leader Education Program Feasibility Trial
Acronym: SPIN-SSLED-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Professor, Faculty of Medicine, McGill University Senior Investigator, Lady Davis Institute for Medical Research, Jewish General Hospital, Lady Davis Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-112
Record Dates: First submitted 2018-04-15; First posted 2018-04-26 (Actual); Results first posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Scleroderma; Systemic Sclerosis
Keywords: Scleroderma; Systemic Sclerosis; Support group; Training; Feasibility
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPIN-SSLED Program (Experimental): 13-session SPIN-SSLED Program
  Interventions: Other: SPIN-SSLED Program

INTERVENTIONS:
Other: SPIN-SSLED Program — The program includes 13 modules that will be delivered live via webinar over the course of the 3-month program. Each module will be delivered in a 60- to 90-minute session. Module topics include (1) the leader's role; (2) starting a support group; (3) structuring a support group meeting; (4) scleroderma 101; (5) successful support group culture; (6 &7) managing support group dynamics I and II; (8) grief and crisis in scleroderma; (9) marketing and recruitment; (10) the continuity of the group; (11) supporting yourself as a leader; (12) virtual support group meetings, (13) support group leader resources. Participants will receive a workbook, be shown filmed vignettes, and will have access to an online resource center.

SUMMARY:
Many people living with a rare disease turn to peer-led support groups to cope with their condition and access educational resources. Systemic sclerosis (SSc), or scleroderma, is a rare autoimmune connective tissue disease where peer-led support groups play an important role. There are currently approximately 200 SSc support groups in Canada and the US, most of which are led by people with SSc. Many SSc patients, however, cannot access support groups. In other cases, support groups are not sustained due to factors that include the burden on group leaders living with a serious, unpredictable disease and limited group leadership skills of some untrained leaders. Our partners from Scleroderma Canada and the Scleroderma Foundation in the US are committed to improving support group accessibility and effectiveness. These organizations maintain a list of active support groups, but currently do not provide training or other resources to groups or their leaders. To address this gap, our team, including investigators and patients from the Scleroderma Patient-centered Intervention Network (SPIN), developed the Scleroderma Support group Leader EDucation (SPIN-SSLED) Program, which is designed to improve support group leader confidence and self-efficacy, reduce burnout, improve emotional well-being, and improve health-related quality of life.

In the planned full-scale randomized controlled trial (RCT) that will follow our feasibility trial, we will evaluate whether the SPIN-SSLED Program is effective in improving SSc support group leaders' self-efficacy for carrying out their leader role (primary) and if it reduces burnout, improves emotional well-being, and improves health-related quality of life (secondary). Thus, the SPIN-SSLED Feasibility Trial answers the following research questions: (1) Is a full-scale SPIN-SSLED RCT feasible? (2) Are adaptations needed to the research design for the planned full-scale RCT? (3) Are there ways to improve the SPIN-SSLED Program for delivery in the planned full-scale RCT based on input of support group leaders who participate in the feasibility trial?

DETAILED DESCRIPTION:
People with rare diseases experience many of the same challenges as those with more common diseases, but also face unique challenges, including gaps in knowledge about their disease and limited treatment and support options. Professionally organized support services are often available for people with more common diseases but are not typically available for people with rare diseases. Instead, many people with rare diseases rely on peer-led support groups for education and to cope with their disease. Support groups may be held face-to-face or online, led by professionals or peers, and have a structured or an unstructured format. Activities typically involve an educational or information-sharing component and the exchange of emotional and practical support.

SSc is a rare, chronic, autoimmune connective tissue disease characterized by abnormal fibrotic processes and excessive collagen production. Peer-led support groups play an important role for people with the disease. There are currently approximately 200 active SSc support groups listed by Scleroderma Canada or the Scleroderma Foundation in the USA, most led by people with the disease. Many people with SSc, however, do not have access to SSc support groups, and many support groups that are initiated are not sustained due to obstacles that could be addressed by providing training to support group leaders. Challenges for patient support group leaders, particularly in rare diseases, include practical difficulties, such as a lack of resources or poor coordination with medical professionals and leader organizations; difficulties with group leadership tasks, such as managing complex group dynamics; and personal challenges, such as managing one's own health condition while supporting others and preventing burnout.

A training and education program could provide the necessary information and skills to improve the ability of SSc peer support group leaders to lead sustainable, effective support groups; reduce their emotional and physical burden; and encourage new leaders to set up support groups where none exist or via the internet. In rare diseases, face-to-face delivery of such a training program is not feasible because current and potential leaders are widely dispersed geographically. Videoconferencing has been used successfully to train educators, health service providers, and parents of children with behavioural difficulties, for example, and is as effective as face-to-face training.

The SPIN-SSLED Program was developed by a team of researchers with expertise in SSc, patient organization representatives, and a Patient Advisory Board comprised of current SSc support group leaders. The program content and design are based on results of our preliminary research on support groups in SSc and informed by instructional material for support group leaders we identified via the internet and by consultations with support group leaders. The program uses a problem-based learning approach. Problem-based learning is a learner-centered approach that integrates theory and practice by providing the necessary knowledge and skills, presenting a complex, real-world problem, then working to identify an approach to solving the problem. To implement this, each module, or learning session, will introduce a topic and provide an overview of key information. Then, there will be a guided discussion among training group participants about possible approaches and solutions. The program includes 13 modules that will be delivered live via webinar over the course of the 3-month program. In addition to the live modules, SPIN-SSLED participants will receive a workbook that summarizes didactic material that is provided and will be shown filmed vignettes demonstrating effective group facilitation techniques and ways to respond to support group issues. SPIN-SSLED participants will also have access to an online resource center that includes a range of helpful tools for leaders including files of SSc related videos to show at meetings and an online forum for leaders to post questions, open only to leaders enrolled in the training program.

The proposed SPIN-SSLED Program Feasibility Trial builds on this background research and will evaluate the feasibility of delivering the SPIN-SSLED Program and of our planned full-scale trial design. The objectives of this study are (1) To evaluate the feasibility of steps needed to take place in the full-scale trial, including the required resources (e.g., staffing, time, and budget), management issues (e.g., related to optimizing performance of personnel and data systems), and scientific aspects (e.g., recruitment of eligible leaders, fidelity of intervention delivery, acceptability of intervention to leaders, assessing performance of outcome measures); (2) To make any necessary modifications to the SPIN-SSLED Program based on participant feedback

The aim of the SPIN-SSLED Feasibility Trial is to collect data related to the study's process, in order to assess the feasibility of the steps that need to take place as part of the main study; required resources (e.g., staffing, time, and budget), management issues (e.g., optimizing performance of personnel and data systems); and scientific aspects (e.g., recruitment rates of eligible leaders, fidelity of intervention delivery, acceptability of intervention to leaders, performance of outcome measures).

Our partners from the Scleroderma Canada and the Scleroderma Foundation will contact group leaders to describe the SPIN-SSLED Feasibility Trial and ascertain interest in participating. SPIN-SSLED personnel will send email invitations with the consent form to interested support group leaders. Following this, support group leaders will be contacted by phone within 48 hours to describe the study, review the consent form, and answer questions assessing eligibility. Eligible patients who verbally accept the offer to enrol in the study will receive an email with the consent form for the study, which they can sign by replying, "I have read the consent form and understand the terms of the feasibility study. I agree to participate in the study testing the feasibility of the SPIN-SSLED Program." We will enroll 10 SSc support group leaders to participate in the program. Based on our previous experience with videoconferencing and consistent with previous trials of videoconference training, to maximize effective interaction and participation, 5 group leaders will be assigned to each training group. Training sessions will be delivered using the GoToMeeting® videoconferencing platform, a high-performance platform that has been used successfully for similar applications.

A survey will be administered to all participants before the trial. The survey will contain a demographics questionnaire designed for this study that includes basic demographic information, such as gender, age and employment status. The survey also includes disease-related variables, such as years since scleroderma diagnosis and questionnaires for all outcome measures. These questionnaires will be administered again upon completion of the program, along with a satisfaction questionnaire. All questionnaires will be completed using the online surveying tool Qualtrics. Once the online survey data is collected, data will be exported to the statistics software program, IBM SPSS.

A description of feasibility outcomes will be presented, including leader eligibility and recruitment, leader enrolment and randomization, technological performance of the videoconferencing system, and treatment fidelity. Qualitative information will inform any necessary changes to the program or trial methods before conducting a full-scale trial. Descriptive statistics will be used to provide means and standard deviations for SPIN-SSLED Program outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Be a current SSc support group leader or have been identified by Scleroderma Canada or the Scleroderma Foundation as a new leader who will initiate a new support group
* Be available to participate at times when sessions are scheduled
* Be English-speaking

Exclusion Criteria:

* Unable to use the internet to access and participate in training sessions or to complete study questionnaires online

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2018-08-10 (Actual); Study Completion 2018-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brett Thombs, PhD, Principal Investigator — Jewish General Hospital and McGill Universit
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Thombs BD, Dyas L, Pepin M, Aguila K, Carrier ME, Tao L, Harb S, Malcarne VL, El-Baalbaki G, Pelaez S, Sauve M, Hudson M, Platt RW; SPIN-SSLED Patient Advisory Team. Scleroderma Patient-centered Intervention Network-Scleroderma Support group Leader EDucation (SPIN-SSLED) program: non-randomised feasibility trial. BMJ Open. 2019 Nov 11;9(11):e029935. doi: 10.1136/bmjopen-2019-029935. PMID 31719073

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Scleroderma Canada and the Scleroderma Foundation were asked to generate a list of 12 interested scleroderma support group leaders. These leaders received an initial email invitation to join the study along with the consent form and the first 10 leaders to consent were enrolled in the study. Participants were recruited from February to March 2018.
Pre-assignment Details: One of the 10 participants who initially indicated that she would participate was hospitalized and was unable to take part before providing informed consent. This participant was replaced with one of the remaining interested support group leaders that were contacted prior to the start of the program. Thus, 10 participants were enrolled.
Period: Overall Study
Arm/Group | SPIN-SSLED Program
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participants can indicate more than one race/ethnicity.
  Participants
    White | 10
    Aboriginal | 1
Relationship status [Count of Participants; unit: Participants]
  Married or living as married | 8
  Separated or divorced | 2
Education [Mean (Standard Deviation); unit: years] | 17.5 (2.7)
Occupational status [Count of Participants; unit: Participants]
  Homemaker | 1
  Part- or full-time employment | 2
  Disability | 3
  Retired | 4
Scleroderma diagnosis [Count of Participants; unit: Participants]
  Limited scleroderma | 4
  Diffuse scleroderma | 5
  Not diagnosed with scleroderma | 1
Years since diagnosis [Mean (Standard Deviation); unit: years] | 10.9 (7.4)
Current leader of scleroderma support group [Count of Participants; unit: Participants] | 10
Years as a support group leader [Mean (Standard Deviation); unit: years] | 3.6 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Participant Feedback on Usability of Program Materials
Description: Participant Interviews. Participants were asked if they found the program to be useful. The number of participants who found the program materials to be useful were recorded
Time Frame: 13 week
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Participant Feedback on Ease of Use of the Go-To Videoconferencing Program
Description: Participant Interviews. Participants were asked if they encountered difficulties during the use of Go-To videoconferencing program. Number of participants who found no difficulty in using the program is reported.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
Participants
  No technical difficulties | 8
  Minor difficulties | 2

3. Primary Outcome: Participant Feedback on Ease of Use of the Online Forum
Description: Participant Interviews. Participants were asked to report the overall technological difficulties that they experienced using the online forum.
Time Frame: 13 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
Participants
  Minimal difficulties | 10
  Other difficulties | 0

4. Primary Outcome: Personnel Requirements
Description: Time logs completed by research staff will be used to assess personnel requirements for the full-scale trial.
Time Frame: 13 weeks
Measure: Number; unit: personnel required
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
personnel required | 0

5. Primary Outcome: Duration of Management of Online Training Group Participation
Description: The challenges related to the management of online training group participation encountered by study personnel, including assisting participants with accessing GoToMeeting and managing Qualtrics for data collection. Time required for management of training groups could not be assigned to individual participants as sometimes the group needed support, and other times an individual did. Thus, the number presented represents the total time required.
Time Frame: 13 weeks
Measure: Number; unit: hours
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
hours | 2

6. Primary Outcome: Percentage of Topics Adequately Covered in the Sessions
Description: Intervention fidelity will be evaluated through the observation of entire sessions for a randomly selected sample of 25% of video-recorded sessions. Raters will evaluate adherence to each session's goals and content using a checklist coding system based on a standardized format. Two raters reviewed 54 topics from 7 randomly chosen modules from both training groups to examine if the contents were adequately covered.
Time Frame: 13 weeks
Measure: Number; unit: percentage
Units Other Than Participants: Topics
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
Number analyzed (Topics) | 54
percentage
  Covered topics | 96
  Not covered topics | 4

7. Primary Outcome: Number of Participants That Reported no Technological Problems
Description: Log of technological problems reported by staff and participants will be maintained and reported descriptively.
Time Frame: 13 weeks
Measure: Number; unit: participants
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
participants
  No technological problems | 8
  Some technological problems | 2

8. Secondary Outcome: The Scleroderma Support Group Leader Self-efficacy Scale (SSGLSS)
Description: The SSGLSS consists of 32 core items that assess the confidence of SSc support group leaders to carry out tasks necessary for leading a support group successfully. Items are scored on a 6-point scale ranging from Strongly Disagree to Strongly Agree (scored 0-5). Possible total scores range from 0 to 160 with higher scores indicating greater self-efficacy.
Time Frame: 13 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
units on a scale | 1.7 [0.67 to 2.72]

9. Secondary Outcome: Personal Health Questionnaire (PHQ-8)
Description: The Personal Health Questionnaire (PHQ-8) is a self-administered 8-item scale to assess depression that has been validated for use in populations with SSc. Items are rated on a 4-point Likert scale (not at all, several days, more than half the days, nearly every day). The total values range from 0 to 24, with higher scores indicating higher levels of depressive symptoms. The difference of pre- and post-trial means was calculated.
Time Frame: baseline and 13 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
score on a scale | 0.38 [-0.50 to 1.27]

10. Secondary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS-29) Profile Version 2.0
Description: The Patient Reported Outcomes Measurement Information System (PROMIS-29) measure contains 29 items, which include four items each for domains reflecting physical function, anxiety, depression, fatigue, sleep disturbance, pain interference, and ability to perform social roles, plus a single item on pain intensity. Total raw scores are obtained by summing item scores for each domain, which are converted into T-scores standardized from the general US population (mean=50, SD=10). High scores represent more of the domain being measured. Thus, on symptom-oriented domains, higher scores represent worse symptomatology. On the function-oriented domains, higher scores represent better functioning.The difference of pre- and post-trial means was calculated.
Time Frame: baseline and 13 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
score on a scale | 0.45 [-0.42 to 1.36]

11. Secondary Outcome: Oldenburg Burnout Inventory (OLBI)
Description: The Oldenburg Burnout Inventory (OLBI) is a 16-item measure of burnout that assesses levels of exhaustion and disengagement in work populations. Items were adapted and reviewed by project investigators for use within the support group leader population. Items are scored on a 4-point scale from 1 (strongly disagree) to 4 (strongly agree). The total values range from 16 to 64, with higher score representing higher level of exhaustion and disengagement. The difference between pre- and post-trial means was calculated.
Time Frame: baseline and 13 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | SPIN-SSLED Program
Number analyzed (Participants) | 10
score on a scale | 0.44 [-0.44 to 1.33]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | SPIN-SSLED Program
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03508661/Prot_SAP_000.pdf